CLINICAL TRIAL: NCT01931059
Title: Acute D2 Receptor Blockade Induced Neuronal Network Changes in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Miklos Argyelan, MD, MD, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13-036
Record Dates: First submitted 2013-08-12; First posted 2013-08-29 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Imaging of the Brain and Antipsychotics; Neuronal Network Changes
Keywords: Imaging; Risperidone; Placebo; antipsychotic
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone then Placebo (Experimental): This group will receive 2 mg (>200lbs), 1.5mg (150-200lbs.) or 1 mg (< 150lbs. of risperidone oral solution on the first day and a placebo on the second day.
  Interventions: Drug: Risperidone; Other: Placebo
- Placebo then Risperidone (Experimental): This group will receive a placebo on the first day and 2mg (> 200lbs.), 1.5mg (150-200lbs), or 1 mg (<150lbs.) of risperidone oral solution on the second day
  Interventions: Drug: Risperidone; Other: Placebo

INTERVENTIONS:
Drug: Risperidone — We gave oral liquid of risperidone one time 1-2 mg depending on subject's weight.
Other: Placebo — We gave oral liquid without active risperidone (pt and provider were both double blinded)

SUMMARY:
To detect the effect of second-generation antipsychotic drug on the neural activity.

DETAILED DESCRIPTION:
To detect functional correlation changes in the brain with anti-psychotic drug administration as compared to placebo, and b.) to measure if these changes correlate with the plasma level of anti-psychotic, and c.) to evaluate if these changes correlate with drug induced symptoms and changes in cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age
* Subject is competent to provide informed consent

Exclusion Criteria:

* Mini Mental Status Exam is less than 28
* Past or current history of any psychotic illness in the subject or in first degree family members
* Self report of illicit drug use (except marijuana) in the past. Use of marijuana during the last 3 month...
* Any use of antipsychotic in the past.
* Any neuro-anatomical lesions on previous brain imaging
* Any use of D2 receptor blocking agent (such as antiemetics) in the last two weeks.
* Any use of any psychotropic medications (SSRI, mood stabilizers, benzodiazepines, stimulants) in the last month.
* MRI contraindications
* Any cardiovascular or cerebrovascular diseases or conditions that predispose patients to hypotension (eg. dehydration, hypovolemia, antihypertensive medication)
* Subjects with diabetes mellitus, metabolic syndrome, hepatic or renal impairment, seizure disorder and any neurological disorder
* QTc interval longer than 450 ms for male and 470 ms for female
* Subjects who used any medications in the last two weeks (to avoid any possible drug-drug interactions)
* Pregnancy
* Individuals who are illiterate and/or visually impaired

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Argyelan, MD, Principal Investigator — Northwell Health
Locations (1):
- Zucker-Hillside Hospital, Glen Oaks, New York, United States

REFERENCES:
- [Background] Ho BC, Andreasen NC, Ziebell S, Pierson R, Magnotta V. Long-term antipsychotic treatment and brain volumes: a longitudinal study of first-episode schizophrenia. Arch Gen Psychiatry. 2011 Feb;68(2):128-37. doi: 10.1001/archgenpsychiatry.2010.199. PMID 21300943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done between 9/4/2013 and 9/19/2014 at the Department of Research at the Zucker Hillside Hospital.
Pre-assignment Details: Subjects were immediately randomized to either Arm 1 or Arm 2.
Groups:
- Risperidone Then Placebo: This group will receive 2 mg (>200lbs), 1.5mg (150-200lbs.) or 1 mg (< 150lbs. of risperidone oral solution on the first day and a placebo on the second day, on third day they did not receive anything.
- Placebo Then Risperidone: This group will receive a placebo on the first day and 2mg (> 200lbs.), 1.5mg (150-200lbs), or 1 mg (<150lbs.) of risperidone oral solution on the second day, on the third day they did not receive anything.
Period: Day 1
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1
Period: Day2
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0
Period: Day3
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Started | 6 | 4
Completed | 5 | 4
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risperidone Then Placebo: This group will receive 2 mg (>200lbs), 1.5mg (150-200lbs.) or 1 mg (< 150lbs. of risperidone oral solution on the first day and a placebo on the second day.
  Risperidone
- Placebo Then Risperidone: This group will receive a placebo on the first day and 2mg (> 200lbs.), 1.5mg (150-200lbs), or 1 mg (<150lbs.) of risperidone oral solution on the second day
  Risperidone
- Total: Total of all reporting groups
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: Because right after enrollment pt inn placebo then risperidone arm was found to be pregnant and was ruled out from the study, no baseline information exist.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 4 | 10
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.4) | 37.5 (10.4) | 34.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject exited study after enrollment due to pregnancy.
  Participants
    Female | 3 | 2 | 5
    Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants] — Population: One subject exited study after enrollment due to pregnancy test came back positive.
  participants
    United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Repeatable Battery for the Assessment of Neuropsychological Status
Description: This will measure the subject's cognitive performance. RBANS is a well-characterized repeatable battery to measure a wide array of cognitive performance in different cognitive domains. We will use Total Score in RBANS: five index scores are computed from the RBANS (immediate memory, language, visuospatial, attention, delayed memory) that are combined to provide the Total Score. The Total Score is expressed as a standardized score normalized to a population mean of 100, with a standard deviation of 15 (possible scores 40-135). Higher scores reflect better performance. More detailed information is available: Randolph C, Tierney MC, Mohr E, Chase TN (June 1998). "The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity". J Clin Exp Neuropsychol. 20 (3): 310-9. doi:10.1076/jcen.20.3.310.823. PMID 9845158.
  Here we calculated the difference of T-scaled total RBANS score between risperidone day and placebo day in all participants
Time Frame: The change of RBANS scores between placebo and treatment conditions on two consecutive days
Measure: Mean (Standard Deviation); unit: RBANS T-Scale point difference
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Number analyzed (Participants) | 6 | 4
RBANS T-Scale point difference | -1.5 (6.6) | -0.5 (7.5)

2. Secondary Outcome: Simpson-Angus Extrapyramidal Side Effects Scale
Description: The secondary outcome measures are the scores from side effect scales (Simpson-Angus Extrapyramidal Side Effects. It will measured in synchrony with Repeated Battery for the Assessment of Neuropsychological Status to explore if any of these measures would correlate with network changes in the brain. The Simpson-Angus scale is 0 if there is no extrapyramidal side effects, and is higher the worst the symptoms are.
Time Frame: 2 times on risperidone day and on placebo day
Population: We analyzed the difference between patients who received drug versus placebo on the first day. 0 would mean no side effects after administration of risperidone or placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Number analyzed (Participants) | 6 | 4
units on a scale | 0 (0) | 0 (0)

3. Other Pre Specified Outcome: Feedback-based Probabilistic Classification Task
Description: On each trial, participants will view one of four images and will be asked to guess whether it belongs to Category A or B. For each participant, the four images will be randomly assigned to be stimuli S1, S2, S3 and S4 (these are abstract visual stimuli denoted with numbers (stiumulus 1, stimulus 2, etc). A different set of similar images (S5-S8; S9-S12, etc) will be used for repeated testing. On any given trial, stimuli S1 and S3 will belong to Category A with 90% probability and to Category B with 10% probability, while stimuli S2 and S4 will belong to Category B with 90% probability and to Category A with 10% probability. Stimuli S1 and S2 will be used in the reward-learning task and S3 and S4 in punishment-learning task. Two stimuli per valence will be employed in order to balance category outcome frequencies, so that one stimulus in each task will be associated with each outcome.
Time Frame: Before every MRI except the 2nd and 4th which will occur during the MRI (5 times - 3 consecutive days)
Population: We lumped individuals from both arms to four groups depending on the task and the medication status and calculated the percentage of correct responses. Due to computer problems 3 subjects' data were lost.
Measure: Mean (Standard Deviation); unit: percentage of correct response
Groups:
- ON - PUNISHMENT: Subject's performance during the peak of the risperidone effect in the punishment part of the task
- OFF - PUNISHMENT: Subject's performance after placebo administration.
- ON - REWARD: Subject's performance during the peak of the risperidone effect in the reward part of the task
- OFF - REWARD: Subject's performance after placebo administration in the reward part of the task
Arm/Group | ON - PUNISHMENT | OFF - PUNISHMENT | ON - REWARD | OFF - REWARD
Number analyzed (Participants) | 7 | 7 | 7 | 7
percentage of correct response | 52.86 (17.99) | 71.43 (21.93) | 61.43 (27.34) | 70.00 (25.17)

ADVERSE EVENTS:
Arm/Group | Risperidone Then Placebo | Placebo Then Risperidone
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No